CLINICAL TRIAL: NCT05339672
Title: Determining the Clinical Relevance of the Interaction Between Enzalutamide and the Opioid Morphine and the DOAC Edoxaban to Improve Rational Pharmacological Care of Patients With Prostate Cancer
Brief Title: Determining the Clinical Relevance of the Interaction Between Enzalutamide and the Opioid Morphine and the DOAC Edoxaban
Acronym: MIND THE GAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MIND THE GAP
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-04

CONDITIONS: Drug-drug Interaction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Morphine: The participating patients are treated with morphine before start of enzalutamide (according to label).
  Interventions: Other: Blood sampling - Pharmacokinetic assessment
- Edoxaban: The participating patients are treated with edoxaban before start of enzalutamide (according to label).
  Interventions: Other: Blood sampling - Pharmacokinetic assessment

INTERVENTIONS:
Other: Blood sampling - Pharmacokinetic assessment — Two pharmacokinetic assessements will be performed (before start of enzalutamide and 4-6 weeks after start of enzalutamide). Each pharmacokinetic assessment consists of 9 samples (3mL blood)

SUMMARY:
Enzalutamide is one of the oncolytic drugs that showed efficacy and safety in most of the features of prostate cancer. Approximately 17% of the patients treated with enzalutamide need pain control. Nearly all opioids are metabolized through one of the CYP enzymes induced by enzalutamide, making optimal pain management difficult. For pain control, while using enzalutamide, morphine is being advised since morphine is mainly glucuronidated by UGT2B7 and to a lesser extent UGT1A1. Enzalutamide is in vitro an inducer of UGT1A1 and may inhibit UGT2B7 which could alter morphine concentrations, though the clinical relevance of this interaction is unknown.

In patients with cancer, Direct Oral Anticoagulants (DOACs) are frequently used since vitamin-K antagonists were reported less effective than DOACs in preventing thromboembolic events. However, DOACs are all metabolized through CYP3A4 or P-gp. Due to interaction potential with DOACs, patients treated with enzalutamide are switched to Low Molecular Weight Heparin (LMWHs) administered subcutaneously which is considered safe but less patient friendly. For patients comfort DOACs are preferred over the use of LMWHs. Since rivaroxaban and apixaban are both major substrates for CYP3A4, combination with enzalutamide is prohibited. Dabigatran is a DOAC which is only metabolized by P-gp and edoxaban is a minor substrate for CYP3A4. Therefore, both might be safe to combine with enzalutamide. However, in patients with an active malignancy edoxaban is preferred according to national guidelines. Still, it is unknown if enzalutamide has a significant effect on the edoxaban exposure.

The purpose of this study is to evaluate the effect of enzalutamide on morphine and edoxaban pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer who will start treatment with enzalutamide within label
* Patients who are on treatment with opioids and/or therapeutic anticoagulation, that are treated with or willing and able to switch to morphine (2 dd extended release equivalent dose) and/or edoxaban (30mg or 60mg OD, according to the label)
* Age at least 18 years
* Patients who are able and willing to give written informed consent prior to screening
* Patients from whom it is possible to collect blood samples
* Life expectancy of > 3 months
* Stable renal function and renal clearance > 50ml/min

Exclusion Criteria:

* Patients who are co-treated with drugs that could interfere with the metabolism of enzalutamide, edoxaban and/or morphine

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer starting enzalutamide therapy
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
To determine the change in morphine and morphine-6-glucuronide exposure | 4-6 weeks after start of enzalutamide
  Change in AUC0-12hr
To determine the change in edoxaban and M4 exposure | 4-6 weeks after start of enzalutamide
  Change in AUC0-24hr

SECONDARY OUTCOMES:
To evaluate the pain control in patients treated with and without enzalutamide and morphine | 4-6 weeks after start of enzalutamide
  Change in Numeric Rating Scale (NRS). The pain NRS is a single 11-point numeric scale, with 0 representing no pain and 10 representing extreme pain.
To evaluate the safety of the combination of enzalutamide with edoxaban and/or morphine | 4-6 weeks after start of enzalutamide
  monitored with CTC-AE v 5.0 criteria.
To evaluate the effect of edoxaban and/or morphine on enzalutamide exposure | 4-6 weeks after start of enzalutamide
  Change in Ctrough of enzalutamide

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboudumc, Nijmegen
  - Franciscus Gasthuis en Vlietland hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: No